CLINICAL TRIAL: NCT01047683
Title: Evaluation of the Efficacy and Safety of AMR101 (Ethyl Icosapentate) in Patients With Fasting Triglyceride Levels ≥ 500 mg/dL and ≤ 2000 mg/dL
Brief Title: Efficacy and Safety of AMR101 (Ethyl Icosapentate) in Patients With Fasting Triglyceride (Tg) Levels ≥ 500 and ≤ 2000 mg/dL
Acronym: MARINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMR-01-01-0016; The MARINE Study (Other: Amarin Pharma Inc.)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; omega-3 fatty acids; statin; triglycerides; lipids; EPA; docosahexaenoic acid; fish; fatty acids; fibrates; niacin; lipid; atorvastatin; Lovaza; simvastatin; lovastatin; pravastatin; fluvastatin; rosuvastatin; Trilipix; Vytorin; Simcor; ezetimibe; Zetia; ethyl-EPA; ethyl icosapentate; Crestor; Zocor; Lipitor; Niaspan; LDL; HDL; cholesterol; dyslipidemia; VASCEPA; icosapent ethyl
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — eicosapentaenoic acid ethyl ester; eicosapentaenoic acid ethanolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AMR101 (ethyl icosapentate) - 2 g/day (Experimental)
  Interventions: Drug: AMR101 (ethyl icosapentate) - 2 g/day
- AMR101 (ethyl icosapentate) - 4 g/day (Experimental)
  Interventions: Drug: AMR101 (ethyl icosapentate) - 4 g/day

INTERVENTIONS:
Drug: AMR101 (ethyl icosapentate) - 4 g/day — AMR101 (ethyl icosapentate) 4 capsules/day for 12 weeks (Weeks 1-12)
  Other Names: VASCEPA® (icosapent ethyl)
  Arms: AMR101 (ethyl icosapentate) - 4 g/day
Drug: AMR101 (ethyl icosapentate) - 2 g/day — AMR101 (ethyl icosapentate) 2 capsules/day with placebo 2 capsules/day for 12 weeks (Weeks 1-12)
  Other Names: VASCEPA® (icosapent ethyl)
  Arms: AMR101 (ethyl icosapentate) - 2 g/day
Drug: Placebo — Placebo 4 capsules/day for 12 weeks (Weeks 1-12)
  Arms: Placebo

SUMMARY:
The primary objective is to determine the efficacy of AMR101 (ethyl icosapentate) compared to placebo in lowering fasting triglyceride levels in patients with very high fasting triglyceride levels ≥ 500 and ≤ 2000 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages >18
* Fasting triglyceride ≥500 mg/dL and ≤2000 mg/dL
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant
* Use of non-statin lipid-altering drugs which cannot be stopped including fibrates, niacin, fish oil and other products containing omega-3 fatty acids or other dietary supplements with potential lipid-altering effects
* History of pancreatitis
* History of bariatric surgery or currently on weight loss drugs
* Uncontrolled hypertension (BP > 160/100)
* HIV infection or on treatment with HIV-protease inhibitors, cyclophosphamide,or isotretinoin
* Consumption of more than 2 alcoholic beverages per day
* History of cancers (except if been disease free for >5 years OR history was basal or squamous cell skin cancer)
* Participation in another clinical trial involving an investigational agent in the last 30 days
* Other parameters will be assessed at the study center to ensure eligibility for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (16):
  - Amarin Investigational Site, Sacramento, California
  - Amarin Investigational Site, Golden, Colorado
  - Amarin Investigational Site, Miami, Florida
  - Amarin Investigational Site, Ocala, Florida
  - Amarin Investigational Site, Addison, Illinois
  - Amarin Investigational Site, Chicago, Illinois
  - Amarin Investigational Site, Louisville, Kentucky
  - Amarin Investigational Site, Butte, Montana
  - Amarin Investigational Site, Raleigh, North Carolina
  - Amarin Investigational Site, Winston-Salem, North Carolina
  - Amarin Investigational Site, Cincinnati, Ohio
  - Amarin Investigational Site, Lyndhurst, Ohio
  - Amarin Investigational Site, Tulsa, Oklahoma
  - Amarin Investigational Site, Corpus Christi, Texas
  - Amarin Investigational Site, Houston, Texas
  - Amarin Investigational Site, Richmond, Virginia
- Denmark (2):
  - Amarin Investigational Site, Aalborg
  - Amarin Investigational Site, Herlev
- Amarin Investigational Site, Oulu, Finland
- Germany (5):
  - Amarin Investigational Site, Dresden
  - Amarin Investigational Site, Giessen
  - Amarin Investigational Site, Magdeburg
  - Amarin Investigational Site, München
  - Amarin Investigational Site, Nuremberg
- India (5):
  - Amarin Investigational Site, Ahmedabad
  - Amarin Investigational Site, Bangalore
  - Amarin Investigational Site, Gopālapuram
  - Amarin Investigational Site, Indore
  - Amarin Investigational Site, Mysore
- Italy (2):
  - Amarin Investigational Site, Genova
  - Amarin Investigational Site, Palermo
- Mexico (3):
  - Amarin Investigational Site, Guadalajara, Jalisco
  - Amarin Investigational Site, Mexico City
  - Amarin Investigational Site, Monterrey Nuevo Leon
- Netherlands (4):
  - Amarin Investigational Site, Amsterdam
  - Amarin Investigational Site, Groningen
  - Amarin Investigational Site, Rotterdam
  - Amarin Investigational Site, Utrecht
- Russia (2):
  - Amarin Investigational Site, Moscow
  - Amarin Investigational Site, Saint Petersburg
- South Africa (6):
  - Amarin Investigational Site, Bloemfontein
  - Amarin Investigational Site, Cape Town
  - Amarin Investigational Site, Johannesburg
  - Amarin Investigational Site, Parktown
  - Amarin Investigational Site, Pretoria
  - Amarin Investigational Site, Somerset West
- Ukraine (4):
  - Amarin Investigational Site, Ivano-Frankivsk
  - Amarin Investigational Site, Kiev
  - Amarin Investigational Site, Kyiv
  - Amarin Investigational Site, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bays HE, Ballantyne CM, Kastelein JJ, Isaacsohn JL, Braeckman RA, Soni PN. Eicosapentaenoic acid ethyl ester (AMR101) therapy in patients with very high triglyceride levels (from the Multi-center, plAcebo-controlled, Randomized, double-blINd, 12-week study with an open-label Extension [MARINE] trial). Am J Cardiol. 2011 Sep 1;108(5):682-90. doi: 10.1016/j.amjcard.2011.04.015. Epub 2011 Jun 16. PMID 21683321
- [Result] Bays HE, Braeckman RA, Ballantyne CM, Kastelein JJ, Otvos JD, Stirtan WG, Soni PN. Icosapent ethyl, a pure EPA omega-3 fatty acid: effects on lipoprotein particle concentration and size in patients with very high triglyceride levels (the MARINE study). J Clin Lipidol. 2012 Nov-Dec;6(6):565-72. doi: 10.1016/j.jacl.2012.07.001. Epub 2012 Jul 24. PMID 23312052
- [Result] Bays HE, Ballantyne CM, Braeckman RA, Stirtan WG, Soni PN. Icosapent ethyl, a pure ethyl ester of eicosapentaenoic acid: effects on circulating markers of inflammation from the MARINE and ANCHOR studies. Am J Cardiovasc Drugs. 2013 Feb;13(1):37-46. doi: 10.1007/s40256-012-0002-3. PMID 23325450
- [Result] Braeckman RA, Manku MS, Bays HE, Stirtan WG, Soni PN. Icosapent ethyl, a pure EPA omega-3 fatty acid: effects on plasma and red blood cell fatty acids in patients with very high triglyceride levels (results from the MARINE study). Prostaglandins Leukot Essent Fatty Acids. 2013 Sep;89(4):195-201. doi: 10.1016/j.plefa.2013.07.005. Epub 2013 Aug 1. PMID 23992935
- [Result] Bays HE, Ballantyne CM, Braeckman RA, Stirtan WG, Doyle RT Jr, Philip S, Soni PN, Juliano RA. Icosapent Ethyl (Eicosapentaenoic Acid Ethyl Ester): Effects Upon High-Sensitivity C-Reactive Protein and Lipid Parameters in Patients With Metabolic Syndrome. Metab Syndr Relat Disord. 2015 Aug;13(6):239-47. doi: 10.1089/met.2014.0137. Epub 2015 Apr 20. PMID 25893544
- [Result] Ballantyne CM, Bays HE, Braeckman RA, Philip S, Stirtan WG, Doyle RT Jr, Soni PN, Juliano RA. Icosapent ethyl (eicosapentaenoic acid ethyl ester): Effects on plasma apolipoprotein C-III levels in patients from the MARINE and ANCHOR studies. J Clin Lipidol. 2016 May-Jun;10(3):635-645.e1. doi: 10.1016/j.jacl.2016.02.008. Epub 2016 Feb 23. PMID 27206952
- [Result] Ballantyne CM, Bays HE, Philip S, Doyle RT Jr, Braeckman RA, Stirtan WG, Soni PN, Juliano RA. Icosapent ethyl (eicosapentaenoic acid ethyl ester): Effects on remnant-like particle cholesterol from the MARINE and ANCHOR studies. Atherosclerosis. 2016 Oct;253:81-87. doi: 10.1016/j.atherosclerosis.2016.08.005. Epub 2016 Aug 20. PMID 27596132
- [Result] Bays HE, Ballantyne CM, Doyle RT Jr, Juliano RA, Philip S. Icosapent ethyl: Eicosapentaenoic acid concentration and triglyceride-lowering effects across clinical studies. Prostaglandins Other Lipid Mediat. 2016 Sep;125:57-64. doi: 10.1016/j.prostaglandins.2016.07.007. Epub 2016 Jul 11. PMID 27418543
- [Result] Mosca L, Ballantyne CM, Bays HE, Guyton JR, Philip S, Doyle RT Jr, Juliano RA. Usefulness of Icosapent Ethyl (Eicosapentaenoic Acid Ethyl Ester) in Women to Lower Triglyceride Levels (Results from the MARINE and ANCHOR Trials). Am J Cardiol. 2017 Feb 1;119(3):397-403. doi: 10.1016/j.amjcard.2016.10.027. Epub 2016 Nov 1. PMID 27939227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day
Started | 76 | 76 | 77
Completed | 71 | 70 | 74
Not Completed | 5 | 6 | 3
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Withdrew Consent | 1 | 4 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Triglycerides >2000 mg/dL | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Total
Number analyzed (Participants) | 76 | 76 | 77 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.34) | 53.4 (9.34) | 51.9 (10.27) | 52.9 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 18 | 54
  Male | 58 | 58 | 59 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 67 | 67 | 202
  Other | 8 | 9 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Triglyceride Lowering Effect
Description: Median percent change from baseline to Week 12 in fasting serum triglyceride levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: Intent-to-treat population: randomized patients who received >= 1 dose of study drug and had baseline and >= 1 postrandomization efficacy measurement. Only patients with non-missing baseline and Week 12 endpoint values were included.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 75
Percent change from baseline | -7.0 [-30.1 to 18.6] | -26.6 [-41.1 to 0.0] | 9.7 [-19.2 to 42.3]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; A standard deviation of 45% in the TG measurements and a significance level of P < 0.01 required a sample size of 69 completed patients per treatment group to provide greater than or equal to 90% power to detect a difference of 30% between AMR101 and placebo in the percentage of change from baseline in the fasting TG levels; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum test — Nonparametric analysis p values were planned using Wilcoxon rank-sum test for each comparison between AMR101 and placebo. Comparisons between AMR101 and placebo were made using a significance level of 0.01 for the primary endpoint; A prespecified step-down testing procedure was used to control Type I error rate using 4 g/day vs placebo then, if significant, 2 g/day vs placebo; Median Difference (Final Values) = -33.1, 95% CI 2-sided [-46.6 to -21.5] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0051, Wilcoxon rank-sum test; Median Difference (Final Values) = -19.7, 95% CI 2-sided [-33.3 to -5.6] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

2. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Very Low-density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum very low-density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 75
Percent change from baseline | 0.0 [-22.5 to 29.2] | -19.5 [-35.7 to 19.6] | 13.7 [-13.5 to 55.3]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0005, Wilcoxon rank-sum test — Nonparametric analysis p values were planned using Wilcoxon rank-sum test for each comparison between AMR101 and placebo. Comparisons between AMR101 and placebo were made using a significance level of 0.05 for secondary and exploratory endpoints; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -28.6, 95% CI 2-sided [-43.4 to -13.9] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.1152, Wilcoxon rank-sum test; Median Difference (Final Values) = -15.3, 95% CI 2-sided [-30.3 to -0.7] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

3. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Lipoprotein-associated Phospholipase A2 Levels
Description: Median percent change from baseline to Week 12 in serum Lipoprotein-associated Phospholipase A2 levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 70 | 73 | 70
Percent change from baseline | -5.1 [-17.1 to 7.1] | -17.1 [-26.2 to -1.7] | -2.4 [-15.9 to 13.5]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0006, Wilcoxon rank-sum test — Nonparametric analysis p values were planned using Wilcoxon rank-sum test for each comparison between AMR101 and placebo. Comparisons between AMR101 and placebo were made using a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -13.6, 95% CI 2-sided [-20.2 to -6.3] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.2367, Wilcoxon rank-sum test; Median Difference (Final Values) = -5.1, 95% CI 2-sided [-12.3 to 2.2] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

4. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Group in Apolipoprotein B Levels
Description: Median in percent change from baseline to Week 12 in serum Apolipoprotein B levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 70 | 75 | 73
Percent change from baseline | 2.1 [-4.7 to 7.6] | -3.8 [-11.9 to 3.8] | 4.3 [-4.5 to 17.5]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0019, Wilcoxon rank-sum test — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -8.5, 95% CI 2-sided [-13.5 to -3.2] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.2367, Wilcoxon rank-sum test; Median Difference (Final Values) = -2.6, 95% CI 2-sided [-7.8 to 1.9] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

5. Other Pre Specified Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Low-density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum low density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 75
Percent change from baseline | -2.5 [-9.8 to 23.5] | -4.5 [-23.3 to 17.2] | -3.0 [-21.3 to 23.3]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.6768, Wilcoxon rank-sum test — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -2.3, 95% CI 2-sided [-12.9 to 8.1] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.3022, Wilcoxon rank-sum test; Median Difference (Final Values) = 5.2, 95% CI 2-sided [-5.4 to 15.6] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

6. Other Pre Specified Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Non-High-Density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum non-high density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 73 | 76 | 75
Percent change from baseline | 0.0 [-9.0 to 14.1] | -7.7 [-21.6 to -0.1] | 7.8 [-4.1 to 26.6]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum test — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -17.7, 95% CI 2-sided [-25.0 to -11.3] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0182, Wilcoxon rank-sum test; Median Difference (Final Values) = -8.1, 95% CI 2-sided [-15.1 to -1.4] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Events were collected by systematic assessment at each study visit.
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day
Serious Adverse Events (participants affected / at risk) | 0/76 | 1/76 | 1/77
Other Adverse Events (participants affected / at risk) | 12/76 | 10/76 | 2/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AMR101 (Ethyl Icosapentate) - 2 g/Day (N=76) | AMR101 (Ethyl Icosapentate) - 4 g/Day (N=77)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AMR101 (Ethyl Icosapentate) - 2 g/Day (N=76) | AMR101 (Ethyl Icosapentate) - 4 g/Day (N=77)
Diarrhea (Gastrointestinal disorders) | 5 | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 5 | 1
Eructation (Gastrointestinal disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are restricted in sharing data until an abstract presentation or publication of the manuscript.